CLINICAL TRIAL: NCT00801645
Title: Effects of Aerobic Exercise Training on Arterial Function and Insulin Resistance Syndrome in Obese Children: A Randomized Controlled Trial
Brief Title: Effects of Exercise on Arterial Function and Insulin Resistance Syndrome in Pre-pubertal Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Nathalie Farpour-Lambert, Head of the Obesity Care Program, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNF 3200B0-103853
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
Keywords: Obesity; Cardiovascular disease; Endothelial function; Blood pressure; Exercise; Physical activity; Metabolic syndrome; Children; Pediatric
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Motor Activity; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese exercise (Experimental)
  Interventions: Behavioral: Exercise
- Obese Control (No Intervention)
- Lean Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Lean Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — The exercise groups engage in aerobic exercise training three 60-minute sessions per week for 12 weeks, in addition of school physical education. Training sessions consist of 30 minutes of aerobic exercise (walking, running, games, swimming), followed by strength training and stretching.
  Other Names: Physical activity
  Arms: Lean Exercise; Obese exercise

SUMMARY:
The main purpose of this project is to investigate the effects of an exercise program on arterial function and cardiovascular diseases risk factors in obese and lean pre-pubertal children. This information will be used to underpin prevention strategies to reduce cardiovascular diseases in overweight youth.

DETAILED DESCRIPTION:
Introduction: cardiovascular diseases (CVD) are the major contributor to the global burden of non-communicable diseases, one third of all global death being attributed to CVD. Childhood obesity poses a major public health problem and there is increasing evidence that foundation of cardiovascular diseases lays early in life in obese children. There is therefore an urgent need to identify effective prevention strategies. Physical activity is recognized as major determinants of cardiovascular health in adults and adolescents however, little is known in young children. The main purpose of this project is to investigate the effects of a 3-month exercise training program on arterial function and cardiovascular diseases risk factors in obese and lean children.

Methods: This is a randomized controlled trial including 4 groups of pre-pubertal children aged 6 to 11 years old: 1) obese exercise, 2) obese control, 3) lean exercise, and 4) lean control. The exercise groups engage in aerobic exercise training three 60-minute sessions per week for 12 weeks, in addition of school physical education. Training sessions consist of 30 minutes of aerobic exercise (walking, running, games, swimming), followed by strength training and stretching. Controls are relatively inactive. After the 3-month intervention, the obese control group engages in an identical 12-week exercise program and the obese exercise group is encouraged to continue for a total of 6 months. Primary measures include: 24-hour ambulatory systolic and diastolic blood pressure; endothelial function and mechanical indices of the brachial and carotid arteries using a B-mode ultrasound imager; central blood pressure and pulse wave velocity by tonometry of aplanation. Other measures include: body composition, physical activity, cardio-respiratory fitness, nutrition, quality of life, and fasting blood lipids, insulin, glucose, markers of vascular function and inflammation. Testing is performed at baseline, 3, 6 and 24 months in obese children and at baseline and 3 months in lean children.

We hypothesize that exercise training will result in improved arterial function, body composition and markers of the metabolic syndrome in obese children. This information will be used to underpin prevention strategies to reduce CVD risk factors in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* obese children: Pre-pubertal (Tanner stage 1), BMI > 97th age- and gender-specific percentile (Kromeyer-Hauschild et al. 2001).
* lean subjects: Pre-pubertal (Tanner stage 1), BMI > 10th and < 90th age- and gender-specific percentile.

Exclusion Criteria:

* being involved in any weight control, physical activity, or behavioral therapy
* familial history of dyslipidemia or essential hypertension
* medications or hormones, which may influence cardiovascular function, body composition, lipid or glucose metabolism
* orthopedic affection limiting physical activity
* genetic disorder or a chronic disease
* following a therapy for psychiatric problems

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2004-08; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Arterial function | 0-3-6-24 months

SECONDARY OUTCOMES:
Body composition | 0-3-6-24 months
Body mass index | 0-3-6-24 months
Cardiorespiratory fitness | 0-3-6-24 months
Physical activity | 0-3-6-24 months
Insulin resistance | 0-3-6-24 months
Blood lipids | 0-3-6-24 months
Biological markers of endothelial function | 0-3-6-24 months
High sensitive C-reactive protein | 0-3-6-24 months
Resting and ambulatory blood pressure | 0-3-6-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beghetti, PD, Study Director — Pediatric Cardiology Unit, Departement of Child and Adolescent, University Hospital, Geneva; Nathalie J Farpour-Lambert, MD, Principal Investigator — Pediatric Cardiology Unit, Department of Child and Adolescent, University Hospital, Geneva
Locations (1):
- Department of Child and Adolescent, University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Maggio AB, Aggoun Y, Martin XE, Marchand LM, Beghetti M, Farpour-Lambert NJ. Long-term follow-up of cardiovascular risk factors after exercise training in obese children. Int J Pediatr Obes. 2011 Jun;6(2-2):e603-10. doi: 10.3109/17477166.2010.530665. Epub 2010 Dec 10. PMID 21142752
- [Derived] Farpour-Lambert NJ, Aggoun Y, Marchand LM, Martin XE, Herrmann FR, Beghetti M. Physical activity reduces systemic blood pressure and improves early markers of atherosclerosis in pre-pubertal obese children. J Am Coll Cardiol. 2009 Dec 15;54(25):2396-406. doi: 10.1016/j.jacc.2009.08.030. PMID 20082930